CLINICAL TRIAL: NCT04867538
Title: Prevalence, Risk Factors, and Complications of Cholelithiasis in Adults With Short Bowel Syndrome
Brief Title: The Cholelithiasis in Adults With Short Bowel Syndrome
Status: Completed | Type: Observational
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Wang Xinying, Professor, Jinling Hospital, China
Other Study IDs: 201502022-12
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Short Bowel Syndrome
Keywords: Short bowel syndrome; Cholelithiasis; Prevalence; Risk factors
MeSH Terms: conditions — Short Bowel Syndrome; Cholelithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — No intervention

SUMMARY:
Short-term studies have shown that patients with short bowel syndrome (SBS) often develop cholestasis or cholelithiasis. In this retrospective cohort study, we aimed to define the incidence, risk factors, and clinical consequences of cholelithiasis in adults with SBS over an extended time period.

DETAILED DESCRIPTION:
However, only limited data are available regarding cholelithiasis in patients with SBS. The prevalence of cholelithiasis in patients with SBS has been reported only in two studies. Furthermore, few studies have focused on identifying the risk factors for cholelithiasis in patients with SBS. Considering the marked improvements in medical care and nutrition support during the last 2 decades, the current incidence and risk factors for cholelithiasis in patients with SBS are unknown.

The aim of the current study was to provide comprehensive, longitudinal, and long-term data on the incidence of symptomatic and asymptomatic cholelithiasis in a cohort of patients with SBS, in order to identify the prevalence, risk factors, and clinical consequences of cholelithiasis in patients with SBS to aid in the development of protective interventions.

ELIGIBILITY:
Inclusion Criteria:

All eligible adults diagnosed with SBS

Exclusion Criteria:

age <18 years; history of cholelithiasis before SBS diagnosis; cholecystectomy; biliary tract obstruction or no abdominal imaging (CT, MRI, or ultrasound) after SBS diagnosis.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: SBS was defined as intestinal malabsorption disorder caused by extensive bowel resection with a remnant small intestine length of <200cm
Sampling Method: Non-Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
the incidence of cholelithiasis in patients with SBS | 2010/1/1-2019/12/31
  the incidence of symptomatic and asymptomatic cholelithiasis in a cohort of patients with SBS
risk factors | 2010/1/1-2019/12/31
  the risk factors of cholelithiasis in patients with SBS
complications | 2010/1/1-2019/12/31
  the clinical consequences of cholelithiasis in patients with SBS

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao X, Zhang L, Wang S, Xiao Y, Song D, Zhou D, Wang X. Prevalence, Risk Factors, and Complications of Cholelithiasis in Adults With Short Bowel Syndrome: A Longitudinal Cohort Study. Front Nutr. 2021 Nov 29;8:762240. doi: 10.3389/fnut.2021.762240. eCollection 2021. PMID 34912839